CLINICAL TRIAL: NCT04446338
Title: Immune Status: Antibodies Against Severe Acute Respiratory Syndrome Coronavirus 2 in a Sample of the Eye Department (University Eye Hospital and Research Institute Tübingen)
Brief Title: Immune Status SARS-CoV-2 in a Sample of a Tertiary Eye Health Centre
Acronym: CovidImmunEye
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Institute of Clinical Chemistry and Pathobiochemistry, Department of Internal Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 292/2020BO2
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-05

CONDITIONS: History of Covid-19, Seroprevalence
Keywords: Seroprevalence; Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Worker: Staff of the Department of Ophthalmology, University Tuebingen, Germany
  Interventions: Diagnostic Test: Antibody Test

INTERVENTIONS:
Diagnostic Test: Antibody Test — Presence and Titer of Anti-Sars-CoV-2 Antbodies

SUMMARY:
A sequential combination of different antibodies test against SARS-CoV-2 is evaluated. The protocol included a rapid test and several ELISA tests within a defined cohort of healthcare workers.

DETAILED DESCRIPTION:
In the current pandemic, the assessment of actual COVID-19 infections plays an important role in the assessment of the risk and progress of the epidemic. Shortly, more and more rapid tests will be available, the aim of which is to be able to obtain a good overview of the immune status of corresponding samples in a timely manner.

Employees in the health sector are faced with additional challenges, not only due to the tightened hygiene regulations. The concern about infecting other people and/or exposing oneself to a relevant health risk is of great importance. A moderate to high transmission risk can be assumed for ophthalmology. In view of older patients and sometimes unavoidable proximity, targeted and reliable diagnostics can offer the potential to reduce the risk potential for the current situation by determining antibodies.

A rapid diagnosis is not yet available outside of clinical studies, especially since deficits in specificity (contact with other coronaviruses) are to be expected. Studies on the serological reaction are not yet available for longer observation periods, but it can be assumed that positive direct detection of IgG (Anti Sars-CV-2-ELISA; Euroimmun) is available at the latest 3 weeks after the onset of symptoms. Without larger and representative analyses, it is currently unclear whether seroconversion is associated with permanent immunity or a lack of it leads to a possible susceptibility to reinfection. A combined test procedure is therefore to be offered to employees within the framework of a random sample.

The query of anamnestic parameters allows the assignment to different groups (CC: past COVID infection, PC: possible infection, N: asymptomatic). The primary goal of the planned study is to provide a first preliminary evaluation of the tests used in the current context.

ELIGIBILITY:
Inclusion Criteria:

* Employees of the health facility described
* voluntary request for testing

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Employee of the Department of Ophthalmology (at a university institution)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence | through study completion, maximum of one year
  Rate of anti-SARS-CoV-2 Antibodies

SECONDARY OUTCOMES:
Agreement of the test results and questionnaire | through study completion, maximum of one year
  Kappa statistics
Positive predictive / negative values of the tests applied | through study completion, maximum of one year

CONTACTS AND LOCATIONS:
Locations (1):
- University Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No